CLINICAL TRIAL: NCT00888511
Title: Concomitant Tarceva® and Irradiation in Patients in Local-regionally Advanced Non-small Cell Lung Cancer. A Phase II Study
Brief Title: Tarceva And Radiotherapy in Locally Advanced Lung Cancer Non-small Cell Lung Cancer
Acronym: TARLAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Olfred Hansen (Other)
Collaborators: Odense University Hospital (Other); Copenhagen University Hospital at Herlev (Other); Rigshospitalet, Denmark (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other); Naestved Hospital (Other)
Responsible Party: Sponsor-Investigator, Olfred Hansen, MD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.02
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer; Non-small cell lung cancer; Tarceva; Radiotherapy; Local-regionally advanced non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Tarceva; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Tarceva — Tarceva 150 mg/day
Radiation: Radiotherapy — 66 Gy/33 F/5 F per week for 5 weeks

SUMMARY:
The trial is a phase II study of daily Tarceva combined with definitive radiotherapy in inoperable locally advanced non small cell lung cancer (stage IIB-IIIB). The objective of the phase II trial is to examine Tarceva concomitant with curatively intended irradiation 66 Gy (2 Gy x 33 F, 5 F per week).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with histologically or cytologically documented diagnosis locally advanced NSCLC stage IIB to IIIB without pleural effusion
* Performance status ≤2 on the ECOG scale
* Serum bilirubin must be ≤1.5 upper limit of normal (ULN)
* ALAT ≤2 x ULN
* Able to comply with study and follow-up procedures
* Patients with reproductive potential must use effective contraception
* Written (signed) informed consent to participate in the study

Exclusion Criteria:

* Any unstable systemic disease (including active infection, unstable angina, congestive heart failure, severe hepatic, renal, or metabolic disease)
* Any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer)
* Inability to take oral medication, or requirement of intravenous alimentation
* Nursing mothers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olfred Hansen, MD, Principal Investigator — Odense University Hospital
Locations (7):
- Denmark (7):
  - Department of Oncology, Aarhus University Hospital, Aarhus
  - Department of Oncology, Rigshospitalet, Copenhagen
  - Department of Oncology, Copenhagen University Hospital at Herlev, Herlev
  - Department of Oncology, Naestved Hospital, Næstved
  - Laboratory of Radiation Physics, Odense
  - Odense University Hospital, Odense
  - Department of Oncology, Vejle Hospital, Vejle

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2007 - November 2013
Groups:
- Concurrent Tarceva and RT in LA-NSCLC: Tarceva: Tarceva 150 mg/day
  Radiotherapy: 66 Gy/33 F/5 F per week for 5 weeks
Period: Overall Study
Arm/Group | Concurrent Tarceva and RT in LA-NSCLC
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Concurrent Tarceva and RT in LA-NSCLC
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 75 [49 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival from registration according to RECIST 1.1
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Concurrent Tarceva and RT in LA-NSCLC
Number analyzed (Participants) | 15
months | 9.4 [1.7 to 68]

2. Secondary Outcome: Toxicity
Time Frame: 3 years
Reporting Status: Not Posted

3. Secondary Outcome: Local Tumor Control by CT-scan
Time Frame: May 2012
Reporting Status: Not Posted

4. Secondary Outcome: Overall Response Rate (CR + PR)
Time Frame: May 2012
Reporting Status: Not Posted

5. Secondary Outcome: Local Tumor Control at 9 Months Evaluated by PET-CT
Time Frame: May 2012
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival
Time Frame: May 2012
Reporting Status: Not Posted

7. Secondary Outcome: Disease Free Survival
Time Frame: May 2012
Reporting Status: Not Posted

8. Secondary Outcome: Late Toxicity
Time Frame: May 2012
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Concurrent Tarceva and RT in LA-NSCLC
All-Cause Mortality (participants affected / at risk) | 15/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent Tarceva and RT in LA-NSCLC (N=15)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No